CLINICAL TRIAL: NCT00798525
Title: Argatroban Versus Lepirudin in Critically Ill Patients - A Randomized Double-blind Trial
Brief Title: Argatroban Versus Lepirudin in Critically Ill Patients
Acronym: ALiCia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Supply of Lepirudin ended on 01. April 2012, thus trial terminated on 31. March 2012
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-003122-28
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Heparin Induced Thrombocytopenia (HIT)
Keywords: thrombocytopenia; Heparin; Lepirudin; Argatroban; critically ill patients
MeSH Terms: conditions — Thrombocytopenia | interventions — argatroban; lepirudin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PR1 (Active Comparator): Patients treated with Argatroban (Argatra®), a direct thrombin inhibitor
  Interventions: Drug: Argatroban
- PR2 (Active Comparator): Patients treated with Lepirudin (Refludan®), a direct thrombin inhibitor
  Interventions: Drug: Lepirudin

INTERVENTIONS:
Drug: Argatroban — Argatra (Argatroban) will be diluted to 0.6 mg/ml and 0.5 µg/kg/min will be administered continuously in patients without liver disfunction. In patients with liver disfunction, defined by a bilirubin of > 4mg/dl, argatroban will be administered as a continuous infusion of 0,25 µg/kg/min with a final concentration of 0,3 mg/ml.
  Other Names: Argatra®; MA number: 62085.00.0
  Arms: PR1
Drug: Lepirudin — Refludan (Lepirudin) will be diluted to a final concentration of 0.1mg/ml and initiated as a continuous infusion of 5µg/kg/h in patients with continuous renal replacement therapy. In patients with moderate renal impairment (Creatinine ≥1,3 mg/dl) a final concentration 0,2 mg/ml of will be used to provide continuous infusion of 10 µg/kg/h. Patients without renal impairment (Creatinine < 1,3 mg/dl) will receive a continuous infusion of 50 µg/kg/h by a final concentration of 1 mg/ml of Lepirudin.
  Other Names: Refludan®; MA number: EU/1/97/035/003
  Arms: PR2

SUMMARY:
The purpose of this study is to test the hypotheses that argatroban significantly increases efficacy and safety of renal replacement therapy measured as life time of haemodialysis filters as compared to lepirudin

DETAILED DESCRIPTION:
Critically ill patients are at increased risk to develop deep vein thrombosis due to immobilisation and/or the underlying disease. Usually, heparin is used for anticoagulation in these patients. However, a serious complication of heparin therapy is heparin-induced thrombocytopenia type II (HIT). HIT is an immune-mediated syndrome caused by antibodies directed against the heparin-PF4-complex, which bind to platelets via the Fc part, thereby activating platelets causing aggregation and hypercoagulability. Thus, with HIT the risk of thrombosis and organ damage paradoxically even increases during heparin administration. HIT is associated with significant morbidity and mortality if unrecognized. Therefore, patients, who develop thrombocytopenia and/or thrombosis during heparin therapy are suspicious for HIT and have to receive alternative anticoagulants2.

The direct thrombin inhibitor lepirudin (Refludan®) is equally effective as heparin in prevention of deep vein thrombosis and lung embolism3. The elimination half life of lepirudin averages 60 min, but in renal failure it may increase up to 48 hours. Critically ill patients often develop acute renal failure requiring continuous renal replacement therapy. Thus, if lepirudin is used in these patients, intensive dose adjustment is necessary to avoid accumulation and severe bleeding. In contrast, effective anticoagulation is needed to prevent clot formation within the extracorporeal circuit, as clotting substantially increases the patients´ risks and costs of therapy.

Argatroban (Argatra®), another direct thrombin inhibitor, has recently been shown to be safe and effective in prevention of deep vein thrombosis in patients with HIT. Interestingly, argatroban is eliminated by hepatic metabolism. Therefore, no initial dose adjustment is necessary in patients with renal failure. Preliminary reports document the feasibility of argatroban for anticoagulation during haemodialysis. Observational data in patients undergoing continuous haemodialysis suggest that life time of filters during argatroban anticoagulation is not limited due to clot formation. Thus, argatroban would be safer and more effective than lepirudin in critically ill patients requiring continuous renal replacement therapy.

Therefore, we propose a prospective randomized double-blinded trial to test the hypotheses that argatroban significantly increases efficacy and safety of renal replacement therapy measured as life time of haemodialysis filters as compared to lepirudin

ELIGIBILITY:
Inclusion Criteria:

* Thrombocytopenia suspicious for HIT with decrease in platelet count >50% from baseline obtained at hospital admission
* 4 T´s score for HIT probability >3 AND/OR positive ELISA for HIT
* Age ≥18 years
* Informed consent (if applicable)

Exclusion Criteria:

* Transient thrombocytopenia due to intraoperative bleeding
* Active bleeding
* Intracranial operations
* Liver dysfunction with spontaneous aPTT> 60 sec.
* History of adverse events or sensitivity against study drugs
* Pregnancy
* Age<18 years
* Preexisting psychiatric/neurologic disorders with long-term inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mean running time of a maximum of two consecutive haemodialysis circuits | seven days starting at time of HIT suspicion

SECONDARY OUTCOMES:
Incidence of bleeding, transfusion requirements, thromboembolic events, anaphylactic reactions, and SUSARs, length of hospital stay, mortality, time till target aPTT | seven days starting at time of HIT suspicion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kienbaum, MD, Principal Investigator — Uniklinik Düsseldorf, Klinik für Anästhesiologie
Locations (1):
- Universitätsklinikum Düsseldorf Klinik für Anästhesiologie, Düsseldorf, Germany

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Beiderlinden M, Werner P, Bahlmann A, Kemper J, Brezina T, Schafer M, Gorlinger K, Seidel H, Kienbaum P, Treschan TA. Monitoring of argatroban and lepirudin anticoagulation in critically ill patients by conventional laboratory parameters and rotational thromboelastometry - a prospectively controlled randomized double-blind clinical trial. BMC Anesthesiol. 2018 Feb 9;18(1):18. doi: 10.1186/s12871-018-0475-y. PMID 29426286
- [Derived] Treschan TA, Schaefer MS, Geib J, Bahlmann A, Brezina T, Werner P, Golla E, Greinacher A, Pannen B, Kindgen-Milles D, Kienbaum P, Beiderlinden M. Argatroban versus Lepirudin in critically ill patients (ALicia): a randomized controlled trial. Crit Care. 2014 Oct 25;18(5):588. doi: 10.1186/s13054-014-0588-8. PMID 25344113